CLINICAL TRIAL: NCT01037335
Title: Local Administration of Morphine for Analgesia After Iliac Bone Graft Harvest
Brief Title: Effect of Local Administration of Morphine for Analgesia After Iliac Bone Graft Harvest
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: The Cleveland Clinic (Other)
Collaborators: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GATA 1 123
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Autogenous Bone Grafts
Keywords: bone graft; pain; chronic
MeSH Terms: conditions — Pain; Bronchiolitis Obliterans Syndrome | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control group (Placebo Comparator): 10 ml normal saline (NS) infiltrated into the harvest site, and 1 ml NS was administered intramuscularly.
  Interventions: Drug: morphine
- intramuscular morphine (Active Comparator): 10 ml NS infiltrated into the harvest site and 5 mg morphine (1 ml) intramuscularly
  Interventions: Drug: morphine
- donor site morphine (Active Comparator): 5 mg morphine (10 ml) infiltrated into the harvest site and 1 ml NS intramuscularly.
  Interventions: Drug: morphine

INTERVENTIONS:
Drug: morphine — Group 1 (control group) was given 10 ml normal saline (NS) infiltrated into the harvest site, and 1 ml NS was administered intramuscularly. Group 2 (intramuscular morphine) was given 10 ml NS infiltrated into the harvest site and 5 mg morphine (1 ml) intramuscularly. Group 3 (donor site morphine) was given 5 mg morphine (10 ml) infiltrated into the harvest site and 1 ml NS intramuscularly.

SUMMARY:
The goal of the current study was to evaluate the analgesic efficacy of low-dose morphine administered to the site of bone graft harvesting in patients undergoing orthopedic surgery. In addition to short-term analgesic effects, the incidence of chronic donor site pain was evaluated 1,3,6 m after surgery.

DETAILED DESCRIPTION:
The protocol is approved by the Institutional Review Board at Gülhane Military Medical Academy Haydarpaşa Training Hospital (Istanbul, Turkey) and written informed consent will be obtained from each patient. Sixty adult patients scheduled to undergo elective upper extremity bone fractures using autogenous bone grafts will be enrolled in this prospective, randomized, double-blind study. Patients were eligible for participation if they were greater than 18 yr of age, they weighed more than 40 kg, they were American Society of Anesthesiologists physical status I or II, and they could operate a patient-controlled analgesia (PCA) device and had no allergies to morphine.

All surgical procedures will be performed using a partial thickness posterior iliac crest bone graft harvested through a lateral oblique incision just cephalad to the crest. Anesthesia was induced with 2 mg/kg propofol and 5 mg/kg fentanyl and maintained with sevoflurane in 50% oxygen in air. After the graft was harvested and hemostasis will be achieved, patients will be randomly assigned to one of three treatment groups using a computer- generated random number table. Group 1 (control group) was given 10 ml normal saline (NS) infiltrated into the harvest site, and 1 ml NS was administered intramuscularly. Group 2 (intramuscular morphine) was given 10 ml NS infiltrated into the harvest site and 5 mg morphine (1 ml) intramuscularly. Group 3 (donor site morphine) was given 5 mg morphine (10 ml) infiltrated into the harvest site and 1 ml NS intramuscularly. All intramuscular injections were administered in the deltoid muscle at the same time as harvest site infiltration. The study medications were prepared by the pharmacy and administered by the surgeon and anesthesiologist, who were blinded to their contents. In the recovery room, patients were connected to a PCA pump (Abbott PCA Plus, Abbott Laboratories, North Chicago, IL) containing 1 mg/ml morphine. The initial settings were an incremental dose of 1.5 ml, a lockout interval of 8 min, and a 4-h limit of 30 ml. The incremental dose was increased to 2.0 ml and the 4-h limit was increased to 45 ml if analgesia was inadequate after 1 h. If analgesia was inadequate after an additional hour, the incremental dose was further increased to 2.5 ml. Patients were asked to quantify their pain from both the donor and the upper extremity surgery incision sites on a verbal analog pain scale of 0-10, with 0 representing no pain and 10 the worst imaginable pain. Pain assessments were made by a blinded research nurse observer 2, 4, 6, 8, 12, and 24 h after completion of surgery. In addition, PCA morphine use was recorded at these six time intervals. Analgesic duration was defined as the time from local administration of study drug to the first requirement of PCA morphine. At 1m, 3 m and 6 m yr after surgery, patients will be interviewed by telephone by a blinded investigator, and a detailed questionnaire similar to that reported in a previous study on donor site pain will be completed. The presence and subjective characteristics of any residual donor site pain, including its quality, severity, and frequency, as well as provoking factors and treatment received, will be recorded.

ELIGIBILITY:
Exclusion Criteria:

* Patients on opioids
* Neuropathic disease
* Chronic conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
pain after procedure | first 24 hrs

SECONDARY OUTCOMES:
chronic pain formation | 1,3 and 6m

CONTACTS AND LOCATIONS:
Overall Officials: alparslan turan, md, Study Director — cleveland Clinic, outcomes research